CLINICAL TRIAL: NCT01801449
Title: A Pilot Open-Label Study of Rilonacept (Arcalyst) in the Deficiency of the Interleukin-1 Receptor Antagonist (DIRA)
Brief Title: Rilonacept for Deficiency of the Interleukin-1 Receptor Antagonist (DIRA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Collaborators: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130086; 13-AR-0086 (Other: The National Institutes of Health)
Record Dates: First submitted 2013-02-27; First posted 2013-02-28 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: DIRA
Keywords: DIRA; Clinical Trial; IL-1; Autoinflammatory Syndrome; Rilonacept
MeSH Terms: interventions — rilonacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rilonacept Treatment (Experimental): Rilonacept loading dose of 4.4 mg/kg/week followed by maintenance dose of 2.2 mg/kg/week. Total duration of the study 24 months. Maintenance dose could be escalated to 4.4 mg/kg/week or further to 6.6 mg/kg/week for 3 months only.
  Interventions: Drug: Rilonacept

INTERVENTIONS:
Drug: Rilonacept

SUMMARY:
Background:

- Deficiency of the IL-1 receptor antagonist (DIRA) is a condition that causes repeated episodes of inflammation. People with DIRA can have rashes, fever, and joint pain. Most treatments for DIRA are intended to control the immune system to stop these inflammations. There are drugs that can treat DIRA, but they have to be given daily as injections. Researchers want to try another drug, rilonacept, as a treatment for DIRA. It needs to be given only once a week. Rilonacept will be given to individuals who are at least 3 months old and who have DIRA.

Objectives:

- To test the safety and effectiveness of rilonacept for children and adults with DIRA.

Eligibility:

- Individuals at least 3 months old who have DIRA.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Other tests to study pain and movement will be given. Imaging studies such as bone density scans and x-rays may also be taken.
* Participants will have a minimum of four to five study visits over 12 months. Those who are on different anti-inflammatory drugs (such as anakinra) will stop taking them before beginning the study visits.
* Participants will have rilonacept injections weekly while on this study. The dose will be adjusted as needed to help treat the DIRA symptoms. Participants will keep a diary to monitor their symptoms and any side effects.
* Treatment with rilonacept will be given for 1 year. Participants will have study visits to monitor the treatment. They will provide blood samples and have other tests at these study visits.

DETAILED DESCRIPTION:
Autoinflammatory diseases are illnesses characterized by episodes of inflammation that, unlike autoimmune disorders, lack the production of high titer autoantibodies or antigen-specific T cells. There is growing genetic and clinical evidence that specific cytokine pathways are dysregulated. Monogenic defects in the IL-1 pathway cause cryopyrin associated periodic syndromes (CAPS) and deficiency of the IL-1 receptor antagonist (DIRA), the latter is caused by mutations affecting the IL-1-receptor antagonist gene (IL1RN). Both disorders respond with complete resolution of the inflammatory response to treatment with the short acting IL-1 blocking agent anakinra. This exploratory study aims to examine the utility of the long acting IL-1 inhibitor rilonacept (rilonacept; Regeneron Pharmaceuticals, Inc.)

This pilot study is designed to address: 1) the utility and dosage of rilonacept needed to achieve inflammatory remission in children with DIRA who have shown a response to treatment with anakinra [Kineret[registered]]; and 2) to evaluate the safety and pharmacokinetics in young children on rilonacept.

Rilonacept is a recombinant fusion protein with picomolar affinity for IL-1 and a half-life of approximately 7.5 days in humans. It is approved by the Food and Drug Administration (FDA) for the treatment of adults and children 12 years of age and older with Cryopyrin-Associated Periodic Syndromes (CAPS), and was tested in the clinically milder forms of CAPS including Familial Cold Autoinflammatory Syndrome (FCAS) and Muckle-Wells Syndrome (MWS).

In this study, clinical, and laboratory parameters will initially be measured at baseline following a withdrawal of anakinra for 24 hours. Subjects will receive a course of therapy with rilonacept that is predicted to induce inflammatory remission. Clinical and laboratory measures of inflammation will be assessed; rilonacept dose escalation will be implemented as necessary to achieve clinical and laboratory remission. Subjects will remain on study for 12 months and primary end point will be evaluated at 6 months.

Those subjects who complete the 1-year treatment period and maintain improved clinical and laboratory parameters compared to baseline values, may continue to receive study medication at their current dose. Principal investigator will help to obtain insurance coverage for rilonacept for their continued treatment, and will discuss with Regeneron Pharmaceuticals, Inc. for additional supplies of rilonacept for these subjects.

ELIGIBILITY:
* INCLUSION CRITERIA

  1. Male or female pediatric and adult subjects with mutation positive IL1RN indicating DIRA. For the first five patients enrolled, they must have been on a stable dose of anakinra during the 2-week period prior to screening visit. If the subject is on other medications such as NSAIDs, methotrexate and/or oral steroids, it is a requirement that these doses have been stable during the 2-week period prior to screening visit.
  2. Subjects greater or equal to 3 months of age (however the first 5 patients enrolled will be over 2 years of age). Subjects 3 months old or older will be enrolled after SMC data review of the first 5 enrolled patients.
  3. Participation in NIH study #03-AR-0173 ( Studies of the Natural History, Pathogenesis and Outcome of Autoinflammatory Diseases (NOMID/CAPS, DIRA, CRMO, Still s Disease, Behcet s Disease, and other Undifferentiated Autoinflammatory Diseases )
  4. Subjects currently treated with anakinra may be enrolled in this study even though their DIRA may be quiescent. For these subjects, a history of active DIRA prior to treatment with anakinra will be sufficient. Subjects will not take anakinra 24 hours before initiation of drug treatment. Treatment naive patients will also be enrolled after SMC data review of the first 5 enrolled patients.
  5. Females of childbearing potential (young women who have had at least one menstrual period regardless of age) must have a negative serum pregnancy test at screening and a urine pregnancy test prior to administration of study medication.
  6. Females of childbearing age and men able to father a child and who are sexually active, who agree to use two forms of effective birth control, including abstinence.
  7. Negative Purified Protein Derivative (PPD) test using 5 T.U. intradermal testing or the QuantiFERON(SqrRoot) - TB Gold test per the Centers for Disease Control and Prevention (CDC) guidelines, and no evidence of active tuberculosis (TB) on chest X-ray.

     Subjects with latent TB (positive PPD or QuantiFERON - TB Gold test) currently treated with adequate therapy for at least one month prior to first dose of study medication may be included. Full prophylaxis regimens will be continued while on the study.

     Subjects who have had active TB in the past with documentation of adequate treatment may be included with strict clinical and radiological follow-up as per current guidelines.

     The Infectious diseases service will be consulted regarding all patients with evidence of TB infection (latent or active, current or history) prior to enrollment, and as appropriate during the study.

     Subjects who have been BCG-vaccinated will also be tested. Interpretation of PPD and QuantiFERON - TB Gold test in BCG recipients will be the same as for subjects who have not received BCG vaccine.

     Guardian/parent able to understand, and complete study-related questionnaires.

     Guardian/parent able and willing to give informed consent and abide with the study procedures.

     EXCLUSION CRITERIA

  <!-- -->

  1. Treatment receiving a live virus vaccine (such as the measles, mumps, and rubella vaccine) during the 3 months prior to baseline visit. No live vaccines will be allowed throughout the course of this study.
  2. Presence of active infections or a history of pulmonary TB infection without documented adequate therapy. Subjects with current active TB, or recent close exposure to an individual with active TB, are excluded from the study. Exceptions include patients with latent TB treated with adequate therapy for at least one month prior to the first dose of study medication, and patients with history of TB with documentation of adequate treatment.
  3. Positive test for, or prior history of, HIV, or Hepatitis B or C.
  4. History of malignancy. Subjects deemed cured of superficial malignancies such as cutaneous basal or squamous cell carcinomas, or in situ cervical cancer may be enrolled.
  5. Known hypersensitivity to Chinese Hamster Ovary cell-derived biological or any components of rilonacept.
  6. Presence of any additional rheumatic disease or significant systemic disease. For example, major chronic infectious/ inflammatory/ immunologic disease (such as inflammatory bowel disease, psoriatic arthritis, spondyloarthropathy, SLE in addition to autoinflammatory disease).
  7. Presence of any of the following laboratory abnormalities at enrollment visit:

     creatinine greater than 1.5xULN

     WBC less than 3.0x103/mm3

     ANC less than 800 cells/mL

     platelet count less than 150,000 mm3

     ALT or AST greater than 2.0x ULN.
  8. Lactating, breastfeeding or pregnant females.
  9. Enrollment in any other investigational treatment study or use of an investigational agent, or has not yet completed at least 4 weeks or 5 half-lives, whichever is longer, since ending another investigational device or drug trial.
  10. Subjects for whom there is concern about compliance with the protocol procedures.
  11. Presence of other severe acute or chronic medical or psychiatric condition, or significant laboratory abnormality requiring further investigation that may cause undue risk for the subject s safety, inhibit protocol participation, or interfere with interpretation of study results, and in the judgment of the Investigator would make the subject inappropriate for entry into this study.
  12. Subjects who have received a DMARDs (except methotrexate) and or TNFblocking agent within 4 half-lives prior to study entry.
  13. Men able to father a child and who are sexually active, who do not agree to use 2 form of effective birth control, including abstinence during the duration of the study an for at least 28 days following the last dose of rilonacept.
  14. Females of childbearing potential (woman greater than 12 or who have had at least 1 menstrual period regardless of age) who are sexually active and who do not agree to use 2 effective methods of birth control, including abstinence during the duration of the study an for at least 28 days following the last dose of rilonacept.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-02-12; Primary Completion 2016-04-28 (Actual); Study Completion 2016-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina A Montealegre, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
NIH Biomedical Translational Research Information System

REFERENCES:
- [Background] Aksentijevich I, Masters SL, Ferguson PJ, Dancey P, Frenkel J, van Royen-Kerkhoff A, Laxer R, Tedgard U, Cowen EW, Pham TH, Booty M, Estes JD, Sandler NG, Plass N, Stone DL, Turner ML, Hill S, Butman JA, Schneider R, Babyn P, El-Shanti HI, Pope E, Barron K, Bing X, Laurence A, Lee CC, Chapelle D, Clarke GI, Ohson K, Nicholson M, Gadina M, Yang B, Korman BD, Gregersen PK, van Hagen PM, Hak AE, Huizing M, Rahman P, Douek DC, Remmers EF, Kastner DL, Goldbach-Mansky R. An autoinflammatory disease with deficiency of the interleukin-1-receptor antagonist. N Engl J Med. 2009 Jun 4;360(23):2426-37. doi: 10.1056/NEJMoa0807865. PMID 19494218
- [Result] Garg M, de Jesus AA, Chapelle D, Dancey P, Herzog R, Rivas-Chacon R, Muskardin TLW, Reed A, Reynolds JC, Goldbach-Mansky R, Sanchez GAM. Rilonacept maintains long-term inflammatory remission in patients with deficiency of the IL-1 receptor antagonist. JCI Insight. 2017 Aug 17;2(16):e94838. doi: 10.1172/jci.insight.94838. eCollection 2017 Aug 17. PMID 28814674
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-AR-0086.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Rilonacept Treatment: Rilonacept loading dose of 4.4 mg/kg/week followed by maintenace dose of 2.2 mg/kg/week.Total duration of the study 24 months.
Period: Overall Study
Arm/Group | Rilonacept Treatment
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Rilonacept Treatment: Rilonacept loading dose of 4.4 mg/kg/week followed by maintenace dose of 2.2 mg/kg/week. Total duration of the study 24 months.
Arm/Group | Rilonacept Treatment
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Secondary Outcome: Height
Description: Antropometric measurements - Height z-score
Time Frame: 24 months after rilonacept initiation
Population: Analysis included all subjects
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Rilonacept Treatment
Number analyzed (Participants) | 6
z-score | -1.22 (0.48)

2. Secondary Outcome: Height
Description: Antropometric measurements - Height z-score
Time Frame: Baseline
Population: Analysis included all subjects
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Rilonacept Treatment
Number analyzed (Participants) | 6
z-score | -1.1 (0.41)

3. Secondary Outcome: Weight
Description: Antropometric measurements - Weight z-score
Time Frame: 24 months after rilonacept initiation
Population: Analysis included all subjects
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Rilonacept Treatment
Number analyzed (Participants) | 6
z-score | -0.48 (0.64)

4. Secondary Outcome: Weight
Description: Antropometric measurements - Weight z-score
Time Frame: Baseline
Population: Analysis included all subjects
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Rilonacept Treatment
Number analyzed (Participants) | 6
z-score | -0.59 (0.62)

5. Secondary Outcome: Childhood Health Assessment Questionnaire (CHAQ)
Description: The Childhood Health Assessment Questionnaire (CHAQ) is a patient self-assessment (or parent assessment) tool for how illness affects ability to function in daily life. Includes overall score, overall pain rating, overall global evaluation, subcategories for dressing and grooming, arising, eating, walking, hygiene, reach, grip, and activities. Measured on scale of 0-3 from 'Without any difficulty' (0) to 'Unable to do' (3). The scores are summed and divided by the number of total categories answered to arrive at a final value.
Time Frame: 24 months after rilonacept initiation
Population: Analysis included all subjects
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rilonacept Treatment
Number analyzed (Participants) | 6
Units on a scale | 0.25 (0.38)

6. Secondary Outcome: Childhood Health Assessment Questionnaire (CHAQ)
Description: as for outcome 5
Time Frame: Baseline
Population: Analysis included all subjects
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rilonacept Treatment
Number analyzed (Participants) | 6
Units on a scale | 0.83 (0.74)

7. Secondary Outcome: Dual-energy X-ray Absorptiometry (DEXA) Scores
Description: Mean z-scores of anteroposterior lumbar (AP) spine were used for comparisons
Time Frame: 12 months after rilonacept initiation
Population: Analysis included all subjects
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Rilonacept Treatment
Number analyzed (Participants) | 6
z-score | -0.12 (1.26)

8. Secondary Outcome: Dual-energy X-ray Absorptiometry (DEXA) Scores
Description: Mean z-scores of anteroposterior lumbar (AP) spine were used for comparisons
Time Frame: Baseline
Population: Analysis included all subjects
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Rilonacept Treatment
Number analyzed (Participants) | 6
z-score | -0.08 (1.23)

9. Secondary Outcome: Pediatric Quality of Life Inventory (PedsQL)
Description: Pediatric Quality of Life Inventory (PedsQL)-assess functional impairment and change in treatment and health-related quality of life respectively. Responses on this scale are transformed into a 0-100 scale, with 0 being the worst value for health-related quality of life and 100 being the best possible value for health-related quality of life.
Time Frame: 24 months after rilonacept initiation
Population: Analysis included all subjects
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rilonacept Treatment
Number analyzed (Participants) | 6
Units on a scale | 90.6 (4.85)

10. Secondary Outcome: Pediatric Quality of Life Inventory (PedsQL)
Description: as for outcome 9
Time Frame: Baseline
Population: Analysis included all subjects
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rilonacept Treatment
Number analyzed (Participants) | 6
Units on a scale | 86.6 (8.51)

11. Primary Outcome: Number of Subjects Who Maintained Inflammatory Remission With Rilonacept
Description: Inflammatory remission criteria remission criteria were defined as meeting all of the following criteria: a diary score of <0.5 (reflecting no fever, skin rash or bone pain), normal acute phase reactants (C-reactive protein (CRP) <0.5 mg/dL), no objective skin rash or radiological evidence of active bone lesions on x-ray.
Time Frame: 6 months
Population: Analysis included all subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Rilonacept Treatment
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Rilonacept Treatment
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rilonacept Treatment (N=6)
Thrombocytosis (Blood and lymphatic system disorders) | 1
Otitis Externa (Ear and labyrinth disorders) | 1
Otitis Media (Ear and labyrinth disorders) | 4
Conjunctivitis allergic (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 2
Pharyngitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 2
Allergy to chemicals (Immune system disorders) | 1
Food allergy (Immune system disorders) | 1
Skin reaction (Immune system disorders) | 1
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 6
Blood creatine phosphokinase increased (Investigations) | 2
C-reactive protein increased (Investigations) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 5
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes